CLINICAL TRIAL: NCT01421225
Title: Closed-Loop Insulin Delivery in Children Less Than 7 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Garry Steil, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00000231
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Closed Loop Insulin Delivery; Diabetes; Type 1 Diabetes; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Insulin Pump Therapy first, then Closed Loop (Active Comparator): Standard therapy day 1, Closed-Loop therapy day 2.
  Interventions: Device: Closed-loop Insulin Pump therapy; Device: Standard Insulin Pump Therapy
- Closed Loop first, then Standard Insulin Pump Therapy (Active Comparator): Closed-loop therapy day 1, standard therapy day 2.
  Interventions: Device: Closed-loop Insulin Pump therapy; Device: Standard Insulin Pump Therapy

INTERVENTIONS:
Device: Closed-loop Insulin Pump therapy — Subjects insulin doses were adjusted based on a proportional-integral-derivative algorithm using the continuous glucose monitor readings from 10 PM - noon.
  Other Names: Continuous glucose monitor and computer-linked insulin pump
Device: Standard Insulin Pump Therapy — Subjects insulin doses followed their usual home routine.
  Other Names: Open-Loop Therapy

SUMMARY:
The investigators are conducting this study to find out whether a new device can control blood sugar levels in children who have Type 1 diabetes. In Type 1 diabetes, children have high blood sugar levels because they do not make enough insulin. The standard treatment is to give insulin either by shots or using an insulin pump. A new device, called closed-loop insulin therapy, uses a continuous glucose monitor (CGMs) linked to an insulin pump by a computer. The CGM will send the sugar levels to a computer which automatically figures out how much insulin to give and then gives that amount of insulin through the insulin pump. It will give the child insulin to bring sugar levels down if they are high, and will give less insulin if the child's blood sugar is getting lower. Earlier research using closed-loop insulin therapy has shown the ability for it to improve diabetes care in adults and older children, but there has been no research of closed-loop insulin therapy in young children. This study will compare children's current insulin therapy with the closed-loop system. The knowledge that the investigators gain from this research will help us to figure out whether closed-loop therapy can work in young children, hopefully leading to better Type 1 diabetes care.

DETAILED DESCRIPTION:
We will perform a randomized cross-over study of semi-closed-loop insulin therapy in children less than 7 years old with type 1 diabetes. Subjects will be admitted to the inpatient clinical research center for 48 hours. They will receive their standard home insulin therapy for one day and semi-closed-loop insulin therapy for the other day.

ELIGIBILITY:
Inclusion Criteria:

* Age < 7 years old
* Type 1 Diabetes (as diagnosed by outpatient endocrinologist) with duration greater than 6 months
* Treated with insulin pump therapy for greater than 6 weeks

Exclusion Criteria:

* Any other chronic medical condition
* Weight below 10 kg as this is the minimal required weight for the amount of blood being drawn

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08-15 (Actual); Study Completion 2013-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dauber, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dauber A, Corcia L, Safer J, Agus MS, Einis S, Steil GM. Closed-loop insulin therapy improves glycemic control in children aged <7 years: a randomized controlled trial. Diabetes Care. 2013 Feb;36(2):222-7. doi: 10.2337/dc12-1079. Epub 2012 Oct 1. PMID 23033237

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Insulin Pump Therapy First: The subjects in this arm received Standard Insulin Pump therapy on day 1 followed by Closed-Loop Insulin therapy on day 2.
  Closed-loop Insulin therapy: Subjects' insulin dose will be adjusted based on a proportional-integral-derivative algorithm using the continuous glucose monitor readings from 10 PM - noon.
  Standard Insulin Pump Therapy: Patients will receive standard insulin pump therapy as per their usual home insulin protocol.
- Closed-Loop Insulin Therapy First: The subjects in this arm receive closed-loop insulin therapy on day 1 followed by standard insulin pump therapy on day 2.
  Closed-loop Insulin therapy: Subjects' insulin dose will be adjusted based on a proportional-integral-derivative algorithm using the continuous glucose monitor readings from 10 PM - noon.
  Standard Insulin Pump Therapy: Patients will receive standard insulin pump therapy as per their usual home insulin protocol.
Period: Overall Study
Arm/Group | Standard Insulin Pump Therapy First | Closed-Loop Insulin Therapy First
Started | 4 | 6
Completed | 4 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Insulin Pump Therapy First | Closed-Loop Insulin Therapy First | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 3.7 (1.3) | 5.5 (0.9) | 5.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Glycemic Control
Description: Time spent within target glucose range based on the glucose meter measurements between 10 PM and 8 AM. The target range is 110-200 mg/dl as this is the American Diabetes Association defined target overnight range for this age group.
Time Frame: Participants will be followed for the duration of the 48 hour protocol.
Measure: Mean (Standard Error); unit: Hours
Groups:
- Standard Insulin Pump Therapy: Subjects will receive standard insulin pump therapy as per their usual home insulin protocol on day 1 or 2.
- Closed-Loop Insulin Therapy: Subjects insulin doses will be adjusted based on a proportional-integral-derivative algorithm using the continuous glucose monitor readings from 10 PM - noon the following day on day 1 or 2.
Arm/Group | Standard Insulin Pump Therapy | Closed-Loop Insulin Therapy
Number analyzed (Participants) | 10 | 10
Hours | 3.2 (0.77) | 5.3 (0.66)
Statistical Analysis 1: Comparison: Standard Insulin Pump Therapy vs Closed-Loop Insulin Therapy; We tested the number of nighttime (10 PM - 8 AM) hours glucose was in the target range (110-200 mg/dL) on each of the two nights for which the patient was followed (one night under Standard Insulin Pump Therapy; one night under Closed-loop Insulin Therapy); Test type: Equivalence — The null hypothesis was that the number of hours would be the same (no effect of control); p = 0.12, t-test, 2 sided — Statistical analysis was performed using a paired t-test; Mean Difference (Final Values) = 2.2

2. Secondary Outcome: Post-prandial Glycemic Control
Description: Peak post-prandial blood sugar between 8 AM and noon
Time Frame: Participants will be followed for the duration of the 48 hour protocol
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Closed-Loop Insulin Therpay: Subjects insulin doses will be adjusted based on a proportional-integral-derivative algorithm using the continuous glucose monitor readings from 10 PM - noon the following day on day 1 or two.
Arm/Group | Standard Insulin Pump Therapy | Closed-Loop Insulin Therpay
Number analyzed (Participants) | 10 | 10
mg/dL | 353 (24) | 367 (23)

3. Secondary Outcome: Number of Interventions for Hypoglycemia
Description: The number of interventions for hypoglycemia between 10 PM - 8 AM.
Time Frame: Participants will be followed for the duration of the 48 hour protocol
Measure: Number; unit: Interventions
Arm/Group | Standard Insulin Pump Therapy | Closed-Loop Insulin Therapy
Number analyzed (Participants) | 10 | 10
Interventions | 4 | 5

4. Secondary Outcome: Pre-lunch Blood Glucose Level
Description: Blood glucose levels were documented at 12 pm just prior to being served lunch.
Time Frame: Participants will be followed for the duration of the 48 hour protocol
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Standard Insulin Pump Therapy | Closed-Loop Insulin Therapy
Number analyzed (Participants) | 10 | 10
mg/dL | 273 (24) | 189 (18)

ADVERSE EVENTS:
Time Frame: Participants will be followed for the duration of the 48 hour protocol.
Arm/Group | Standard Insulin Pump Therapy | Closed-Loop Insulin Therapy
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Insulin Pump Therapy (N=10) | Closed-Loop Insulin Therapy (N=10)
Medication Error (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — One episode where mealtime insulin was not administered due to a nursing error. The patient was transiently hyperglycemic until an additional dose of insulin was given. This was a minor event but was unexpected. No harm came to the patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes